CLINICAL TRIAL: NCT01128582
Title: Effect of Rozerem on the Perception of Gastroesophageal Reflux Disease (GERD) Symptoms in Patients With Chronic Insomnia.
Brief Title: Effect of Rozerem on the Perception of GERD Symptoms in Patients With Chronic Insomnia.
Acronym: Rozerem
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southern Arizona VA Health Care System (U.S. Federal Agency)
Responsible Party: Ronnie Fass MD, Southern Arizona VA Health Care System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Rozerem
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-03

CONDITIONS: Gastroesophageal Reflux Disease; Chronic Insomnia
Keywords: GERD; Insomnia; Acid Reflux; Heartburn
MeSH Terms: conditions — Gastroesophageal Reflux; Sleep Initiation and Maintenance Disorders; Heartburn | interventions — ramelteon; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rozerem (Active Comparator): Comparing the effect of Rozerem vs. placebo on GERD symptomatology.
  Interventions: Drug: Rozerem (ramelteon)
- placebo (Placebo Comparator): Comparing the effect of Rozerem vs. placebo on GERD symptomatology
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Rozerem (ramelteon) — dosage= take 1 tablet(8 MG) 20 min. before bedtime
  Other Names: Rozerem; ramelteon
  Arms: Rozerem
Drug: placebo — Comparing the effect of Rozerem vs. placebo on GERD symptomatology.
  Other Names: sugar pill
  Arms: placebo

SUMMARY:
To determine if administration of Rozerem in comparison to a placebo reduces or eliminates gastroesophageal reflux disease(GERD) symptoms in individuals with both GERD and chronic insomnia.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind parallel group study comparing the effect of Rozerem vs. placebo on gastroesophageal reflux disease(GERD) symptomatology as the primary outcome, and sleep quality and quality of life as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Stop H2 blockers 72 hrs prior to starting study
* Stop PPI - 3 weeks prior to staring study
* Heartburn 3+ times a week
* Insomnia 3+ times a week for 3 months
* Erosive esophagitis or Abnormal pH test

Exclusion Criteria:

* On PPI or H2 blocker & not willing to get off
* Normal EGD (upper endoscopy) w/ normal pH test
* Upper Endoscopy(EGD)with erosive esophagitis(EE)- (LA C&D) LA=Los Angeles criteria. Grades include A-D
* Previous gastrointestinal Surgery
* HX of Diabetes/neuropathy
* HX of seizures
* Known psychological abnormalities(depression,anxiety...)
* Clinically Significant Underlying co morbidity
* Narcotic medications(pain meds)
* Regularly taking sleeping medications (2 week wash-out allowed)
* Taking medications that alter sleep-Psychotropic's, antihistamines, Narcotics and Benzodiazepines Sleep Apnea or other sleep disorders-PLM, RLS etc.

Max Age: 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The effect of Rozerem vs. placebo on gastroesophageal reflux disease(GERD) symptomatology. | 4 week trial
  The effect of Rozerem vs. placebo on GERD symptomatology as the primary outcome, and sleep quality and quality of life as secondary outcomes.

SECONDARY OUTCOMES:
Improving quality of sleep and quality of life. | 4 week trial period
  It is believed that poor quality of sleep can cause more esophageal acid exposure. Thus, it is possible that treatment of insomnia may have a beneficial effect on GERD symptomatology as well as actually reduce esophageal acid reflux.

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Fass, MD, Principal Investigator — Southern Arizona Veterans Health Care System-BREFSA
Locations (1):
- Southern Arizona Veterans Health Care System, Tucson, Arizona, United States

REFERENCES:
- [Derived] Jha LK, Fass R, Gadam R, Maradey-Romero C, Nasrollah L, Hershcovici T, Quan SF, Dickman R. The Effect of Ramelteon on Heartburn Symptoms of Patients With Gastroesophageal Reflux Disease and Chronic Insomnia: A Pilot Study. J Clin Gastroenterol. 2016 Feb;50(2):e19-24. doi: 10.1097/MCG.0000000000000322. PMID 25887111